CLINICAL TRIAL: NCT03036293
Title: International Multicenter, Double-blind, Randomized Placebo-controlled Phase IV Clinical Trial of Different Dosing Regimens of Tenoten® in the Treatment of Anxiety in Patients With Somatoform, Stress-related and Other Neurotic Disorders
Brief Title: Tenoten® in the Treatment of Somatoform, Stress-related and Other Neurotic Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-TN-001
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2019-08

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — tenoten

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tenoten, 2 tablets twice daily (4 tablets/day) (Experimental): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets twice daily (4 tablets/day). The tablets should be held in the mouth until dissolution, without meal.
  Interventions: Drug: Tenoten
- Placebo, 2 tablets twice daily (4 tablets/day) (Placebo Comparator): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets twice daily (4 tablets/day). The tablets should be held in the mouth until dissolution, without meal.
  Interventions: Drug: Placebo
- Tenoten, 2 tablets 4 times daily (8 tablets/day) (Experimental): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets 4 times daily (8 tablets/days). The tablets should be held in the mouth until dissolution, without meal.
  Interventions: Drug: Tenoten
- Placebo, 2 tablets 4 times daily (8 tablets/day) (Placebo Comparator): Tablet for oral use. Dose per administration: 2 tablets. 2 tablets 4 times daily (8 tablets/days). The tablets should be held in the mouth until dissolution, without meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenoten — Tablet for oral use.
  Arms: Tenoten, 2 tablets 4 times daily (8 tablets/day); Tenoten, 2 tablets twice daily (4 tablets/day)
Drug: Placebo — Tablet for oral use.
  Arms: Placebo, 2 tablets 4 times daily (8 tablets/day); Placebo, 2 tablets twice daily (4 tablets/day)

SUMMARY:
The purposes of this study are:

* To further examine the efficacy and safety of Tenoten® in the treatment of anxiety in patients with somatoform, stress-related and other neurotic disorders.
* To compare the efficacy of two dosing regimens of Tenoten® (4 tablets daily vs.8 tablets daily, both for 12 weeks) in the treatment of anxiety in patients with somatoform, stress-related and other neurotic disorders.

DETAILED DESCRIPTION:
Design: an international, a multicenter, double-blind, randomized, parallel group placebo-controlled trial to evaluate efficacy and safety of study treatment.

The study will enroll outpatient subjects of both genders aged 18-45 years with verified diagnoses of somatoform, stress-related and other neurotic disorders (F43, F45, F48) and signs of clinically relevant anxiety according to The Hospital Anxiety and Depression scale (HADS).

After signing the informed consent form to participate in the clinical study the subject will be interviewed (complaints, medical history, concomitant therapy) and objective examination will be performed; the subject will fill HADS scale. The severity of anxiety at screening should be ≥ 11 according to HADS. If the subject meets inclusion criteria and has no exclusion criteria he/she will be enrolled into the study. The investigator will determine the severity of anxiety using НАМ-А scale; the subject will fill EQ-5D-3L questionnaire. At Visit 1 (Day 1) the subject will be randomized into one of the treatment groups:

* Group 1: Tenoten® at 2 tablets twice daily (4 tablets/day);
* Group 2: Placebo at 2 tablets twice daily (4 tablets/day);
* Group 3: Tenoten® at 2 tablets 4 daily (8 tablets/day).
* Group 4: Placebo at 2 tablets 4 daily (8 tablets/day). The first dose should be administered at Visit 1 after the visit procedures are completed. Further administration of the study product will be made according to the dosing scheme. The subject will administer the study product and will be followed for 12 weeks during which additional three visits will be made. At Visit 2 (Week 4), Visit 3 (Week 8) and Visit 4 (Week 12) the physician will record patients' complaints and physical examination data, fill HAM-A scale, check the study and concomitant therapy, assess treatment safety and patient compliance with the study treatment. At the final Visit 4 the subject will fill EQ-5D-3L questionnaire and the investigator will fill the Clinical Global Impression Scale Efficacy Index (CGI-EI).

Subjects will be allowed to take symptomatic therapy and medications for their co-morbidities during the study, except for the medicines listed in "Prohibited therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 18-45 years (inclusive).
2. Patients diagnosed with somatoform, stress-related, and other neurotic disorders (F43, F45, and F48), in accordance with the ICD-10 criteria.
3. A moderate and severe anxiety (HADS score ≥ 11) documented at screening.
4. Patients providing signed Informed Consent form for participation in the clinical trial.
5. Patients of reproductive age (of both sexes) using contraceptives and contraceptive methods during the study and for 30 days after the end of participation in the trial.

Exclusion Criteria:

1. Moderate and severe depression symptoms recorded at screening (HADS score ≥ 11).
2. Organic, including symptomatic, mental disorders (F00-09).
3. Mental and behavioural disorders due to psychoactive substance use (F10-19).
4. Schizophrenia, schizotypal and delusional disorders (F20-29).
5. Mood [affective] disorders(F30-39).
6. Phobic (F40) and other anxiety disorders (F41), obsessive-compulsive disorder (F42), dissociative [conversion] disorders (F44), depersonalization-derealization syndrome (F48.1).
7. Behavioral syndromes associated with physiological disturbances and physical factors (F50-59).
8. Disorders of adult personality and behavior (F60-69).
9. Intellectual disabilities (F70-79).
10. Inflammatory and traumatic brain injuries with permanent neurological deficit.
11. Prior diagnosis of a class III or IV cardiovascular disease (according to the New York Heart Association, 1964)
12. Malignant neoplasms/suspected malignant neoplasms.
13. An allergy/intolerance to any of the components of medications used in the treatment.
14. Malabsorption syndrome (including hereditary or acquired lactase or other disaccharidase deficiency) and galactosemia.
15. Any conditions that, from investigator's point of view, may affect the patient's ability to participate in the trial.
16. Hospitalizations or surgeries scheduled for any date during the participation in the study.
17. Patients who, from investigator's point of view, will fail to comply with the observation requirements of the trial or with the dosing regimen of the study drugs.
18. Use of drugs listed in "Prohibited therapy" within a month prior to enrollment.
19. Drug addiction, alcohol use in the amount over 2 units of alcohol a day.
20. Pregnant or breast-feeding women.
21. Participation in other clinical trials within 3 month prior to the enrollment in this study.
22. Patients are related to the research personnel of the investigative site who are directly involved in the trial, or patients who are the immediate family member of the researcher. The 'immediate family member' includes husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
23. Patients working for OOO "NPF "MATERIA MEDICA HOLDING", i.e. the company's employee, temporary contract worker, or appointed official responsible for carrying out the research (or the immediate relative).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Parfenov, DrMedSci, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (22):
- Kazakhstan (2):
  - Kazakh National Medical University named after S.D. Asfendiyarov, Almaty
  - South - Kazakhstan State Pharmaceutical Academy, Shymkent
- Russia (20):
  - Municipal Autonomous Healthcare Institution Order of the Red Banner of Labor City Clinical Hospital No. 1, Chelyabinsk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - The State Autonomic Health Care institution "Interregional clinical and diagnostical center", Kazan'
  - LLC "City Center for Neurology and Pain Management", Kazan'
  - Limited Liability Company "Family policlinic no. 4", Korolyov
  - State Budget Health Care institution of Moscow the City "Scientific and practical psychoneurological center n.a. Z.P. Solovyov" of the Administration of Health Care of Moscow City, Moscow
  - The State Budget Health Care institution of Moscow the City "City clinical hospital No. 12 of the Administration of Health Care of Moscow City", Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - The State Budget Educational institution of High Professional Training I.M. Sechenov First Moscow State Medical University of Ministry of Health Care of the Russian Federation, Hospital of nervous diseases A.Y. Kozhevnikov, Moscow
  - State budgetary institution of public health services of the Nizhniy Novgorod region "Nizhegorod Regional Clinical Hospital named after NA Semashko", Nizhny Novgorod
  - LLC "City Neurological Center" Sibneyromed ", Novosibirsk
  - Pavlov First Saint Petersburg State Medical University/Department of Neurology and Manual Medicine, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University/Department of Neurology with Clinic, Saint Petersburg
  - State-Funded Healthcare Institution of the Samara Region "Samara City N.I. Pirogov Clinical Hospital №1", Samara
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - The State Budget Educational institution of High Professional Training Smolensk State Medical University of Ministry of Health Care of the Russian Federation, Smolensk regional clinical hospital, Smolensk
  - The state budgetary health care institution of the Vladimir region "Regional Clinical Hospital", Vladimir
  - Volgograd State Medical University, Volgograd
  - State Institution of Health of the Yaroslavl Region Clinical Hospital No. 8, Yaroslavl
  - The State Health Care Institution Yaroslavl region "Clinical Hospital №8, Yaroslavl

REFERENCES:
- [Derived] Parfenov VA, Kamchatnov PR, Khasanova DR, Bogdanov EI, Lokshtanova TM, Amelin AV, Maslova NN, Pizova NV, Belskaya GN, Barantsevich ER, Duchshanova GA, Kamenova SU, Kolokolov OV, Glazunov AB. The randomized clinical trial results of the anxiety treatment in patients with somatoform dysfunction and neurotic disorders. Sci Rep. 2021 Dec 20;11(1):24282. doi: 10.1038/s41598-021-03727-5. PMID 34930979 (Retraction: PMID 36104393 Sci Rep. 2022 Sep 14;12(1):15416)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Placebo, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo, 2 Tablets 4 Times Daily (8 Tablets/Day)
Started | 127 | 67 | 131 | 65
Completed | 126 | 64 | 130 | 64
Not Completed | 1 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Placebo, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo, 2 Tablets 4 Times Daily (8 Tablets/Day) | Total
Number analyzed (Participants) | 127 | 67 | 131 | 65 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 127 | 67 | 131 | 65 | 390
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (7.1) | 34.2 (7.4) | 32.8 (7.6) | 34.8 (8) | 33.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 50 | 102 | 52 | 303
  Male | 28 | 17 | 29 | 13 | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kazakhstan | 6 | 6 | 9 | 2 | 23
  Russia | 121 | 61 | 122 | 63 | 367
HAM-A scale baseline score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A). Personality questionnaire designed to identify constitutive anxiety and situational anxiety. The scale consists of 14 items and measures both psychic anxiety and somatic anxiety. Total score is in range 0-56. Includes the symptoms of anxious mood, phobic, emotional, sleep disorders, depressive mood, somatic symptoms - muscular, sensory, cardiovascular, respiratory, gastrointestinal, genitourinary, neurovegetative.
  Anxiety scoring:
  ≤13 - no anxiety; 14-17 - mild anxiety disorder; 18-24 - moderate anxiety disorder;
  ≥25 - severe anxiety.
  units on a scale | 18.84 (5.81) | 17.69 (5.1) | 18.53 (4.32) | 18.2 (6.02) | 18.43 (5.32)
EQ-5D-3L baseline score [Mean (Standard Deviation); unit: units on a scale] — EQ-5D-3L questionnaire (European Quality of Life Instrument). Raw score range 5-15. The lower the better.
  units on a scale | 7.44 (1.44) | 7.51 (1.13) | 7.42 (1.05) | 7.47 (1.45) | 7.45 (1.19)
Hospital Anxiety and Depression Scale (HADS)-Anxiety [Mean (Standard Deviation); unit: units on a scale] — Hospital Anxiety and Depression Scale - Anxiety subscale. Total score 0-21. The lower the better.
  units on a scale | 13.52 (1.79) | 13.01 (1.6) | 13.49 (1.79) | 13.46 (1.99) | 13.41 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean HAM-A Score at 12 Weeks of Treatment: 1. Group 1 (Tenoten®, 4 Tablets a Day); 2. Group 3 (Tenoten®, 8 Tablets a Day).
Description: The Hamilton Anxiety Rating Scale (HAM-A). Personality questionnaire designed to identify constitutive anxiety and situational anxiety. The scale consists of 14 items and measures both psychic anxiety and somatic anxiety. Total score is in range 0-56. Includes the symptoms of anxious mood, phobic, emotional, sleep disorders, depressive mood, somatic symptoms - muscular (pain, convulsions, etc.), sensory (e.g. tinnitus), cardiovascular, respiratory, gastrointestinal, genitourinary, neurovegetative. Major role belongs to behaviour during this interview.
  Anxiety scoring:
  ≤13 - no anxiety; 14-17 - mild anxiety disorder; 18-24 - moderate anxiety disorder;
  ≥25 - severe anxiety.
  Higher values represent a worse outcome
Time Frame: 12 weeks
Population: Raw data from groups placebo-2 and placebo-4 was pooled into combined Placebo group. In accordance with study protocol no dose dependency in placebo effect was assumed. In accordance with study protocol no regiment dependency in placebo effect was assumed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo-2 + Placebo-4: Placebo-2 (2 tablets twice daily) and Placebo-4 (2 tablets 4 times daily)
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
score on a scale
  Week 0 | 18.81 (5.81) | 18.38 (4.32) | 17.88 (5.42)
  Week 12 | 7.26 (4.63) | 6.40 (4.02) | 8.48 (5.13)
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p = 0.0055, ANCOVA; Baseline score used as covariate; Mean Difference (Final Values) = 1.56, 98.33% CI 2-sided [0.217 to 2.91]
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p < 0.0001, ANCOVA; Baseline score used as covariate. Yeo-Johnson transformation with λ=1,09 was applied. Statistical inference performed for transformed values; Mean Difference (Final Values) = 2.56, 98.33% CI 2-sided [1.1 to 3.96] — estimate and CL are backtransformed
Statistical Analysis 3: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day); Mean score differences (begin-end) were compared; Test type: Equivalence — equivalence limits were prespecified as [-2.763; 2.763]; p = 0.0008, ANCOVA; Baseline score used as covariate; Mean Difference (Net) = 0.89, 98.33% CI 2-sided [-0.64 to 2.33]

2. Secondary Outcome: Change From Baseline in the Mean HAM-A Score at 4 Weeks of Treatment: 1.1. Group 1 (Tenoten®, 4 Tablets a Day); 1.2. Group 3 (Tenoten®, 8 Tablets a Day).
Description: as for outcome 1
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
score on a scale
  Week 0 | 18.81 (5.81) | 18.38 (4.32) | 17.88 (5.42)
  Week 4 | 13.73 (5.35) | 13.31 (4.7) | 13.85 (5.34)
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p = 0.08, ANCOVA; Baseline score used as covariate; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.08 to 1.54]
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p = 0.044, ANCOVA; Baseline score used as covariate; Mean Difference (Net) = 0.76, 95% CI 2-sided [0.02 to 1.66]

3. Secondary Outcome: The Mean HAM-A Score at 8 Weeks of Treatment: 2.1. Group 1 (Tenoten®, 4 Tablets a Day); 2.2. Group 3 (Tenoten®, 8 Tablets a Day).
Description: as for outcome 1
Time Frame: 8 weeks
Population: Raw data from groгps placebo-2 and placebo-4 was pooled into combined Placebo group. In accordance with study protocol no dose dependency in placebo effect was assumed. In accordance with study protocol no regiment dependency in placebo effect was assumed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
score on a scale
  Week 0 | 18.81 (5.81) | 18.38 (4.32) | 17.88 (5.42)
  Week 8 | 10.61 (5.44) | 9.88 (4.93) | 10.81 (5.16)
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p = 0.21, ANCOVA; Baseline score used as covariate; Mean Difference (Net) = 0.69, 95% CI 2-sided [-0.4 to 1.78]
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Mean score differences (begin-end) were compared; Test type: Superiority; p = 0.027, ANCOVA; Baseline score used as covariate; Mean Difference (Net) = 1.19, 95% CI 2-sided [0.14 to 2.26]

4. Secondary Outcome: Percentage of Patients Had at Least a 50% Improvement in the HAM-A Score: 3.1. Group 1 (Tenoten® 4 Tablets a Day): After 4, 8 and 12 Weeks; 3.2. Group 3 (Tenoten® 8 Tablets a Day): After 4, 8 and 12 Weeks.
Description: as for outcome 1
Time Frame: 4,8,12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
Participants
  Week 4 | 16 | 18 | 14
  Week 8 | 44 | 55 | 45
  Week 12 | 88 | 96 | 69
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Common OR of event analysis; Test type: Superiority; p = 0.065, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.98 to 1.89] — Bigger OR is better
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Common OR of event analysis; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.22 to 2.33] — Bigger OR is better
Statistical Analysis 3: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 4 frequencies comparison; Test type: Superiority; p = 0.7, Fisher Exact
Statistical Analysis 4: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 8 frequencies comparison; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 5: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 12 frequencies comparison; Test type: Superiority; p = 0.01, Fisher Exact
Statistical Analysis 6: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 4 frequencies comparison; Test type: Superiority; p = 0.57, Fisher Exact
Statistical Analysis 7: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 8 frequencies comparison; Test type: Superiority; p = 0.25, Fisher Exact
Statistical Analysis 8: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 12 frequencies comparison; Test type: Superiority; p = 0.001, Fisher Exact

5. Secondary Outcome: Percentage of Patients With no Anxiety (HAM-A Score <14) in: 4.1. Group 1 (Tenoten®, 4 Tablets a Day); After 4, 8 and 12 Weeks; 4.3. Group 3 (Tenoten®, 4 Tablets a Day); After 4, 8 and 12 Weeks.
Description: as for outcome 1
Time Frame: 4,8,12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
Participants
  Week 4 | 58 | 63 | 66
  Week 8 | 91 | 105 | 96
  Week 12 | 111 | 125 | 111
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Common OR of event analysis; Test type: Superiority; p = 0.46, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.64 to 1.23] — Bigger OR is better
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Common OR of event analysis; Test type: Superiority; p = 0.17, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.9 to 1.79] — Bigger OR is better
Statistical Analysis 3: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 4 frequencies comparison; Test type: Superiority; p = 0.38, Fisher Exact
Statistical Analysis 4: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 8 frequencies comparison; Test type: Superiority; p = 0.67, Fisher Exact
Statistical Analysis 5: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Week 12 frequencies comparison; Test type: Superiority; p = 0.85, Fisher Exact
Statistical Analysis 6: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 4 frequencies comparison; Test type: Superiority; p = 0.71, Fisher Exact
Statistical Analysis 7: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 8 frequencies comparison; Test type: Superiority; p = 0.29, Fisher Exact
Statistical Analysis 8: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Week 12 frequencies comparison; Test type: Superiority; p = 0.007, Fisher Exact

6. Secondary Outcome: Change From Baseline in the Total EQ-5D-3L Score at 12 Weeks of Treatment in Patients From: 5.1. Group 1 (Tenoten®, 4 Tablets a Day); 5.2. Group 3 (Tenoten®, 8 Tablets a Day).
Description: European Quality of Life Instrument questionnaire (EQ-5D-3L) is designed for the evaluation of the quality of life.The score ranges between 5-15. Higher values represent a worse outcome.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
score on a scale
  Week 0 | 7.44 (1.44) | 7.42 (1.05) | 7.48 (1.28)
  Week 12 | 5.84 (1.05) | 5.71 (0.82) | 6.05 (1.07)
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Median changes (begin-end) within groups are compared; Test type: Superiority; p = 0.314, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.00002, 95% CI 2-sided [-0.00002 to 0.33] — Hodges-Lehmann estimator for location difference provided
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Median changes (begin-end) within groups are compared; Test type: Superiority; p = 0.031, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI 2-sided [0 to 1] — Hodges-Lehmann estimator for location difference provided

7. Secondary Outcome: Total CGI Scores in Patients From: 6.1. Group 1 (Tenoten®, 4 Tablets a Day); 6.2. Group 3 (Tenoten®, 8 Tablets a Day).
Description: Clinical Global Impession (CGI) provides a brief assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. Total range 0-16. Higher values represent a worse outcome
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
Number analyzed (Participants) | 126 | 130 | 128
score on a scale | 4.53 (3.21) | 4.55 (2.91) | 5.71 (3.28)
Statistical Analysis 1: Comparison: Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) vs Placebo-2 + Placebo-4; Test type: Superiority; p = 0.0021, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.00001, 95% CI 2-sided [-3 to -0.00001] — Lower is better
Statistical Analysis 2: Comparison: Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) vs Placebo-2 + Placebo-4; Test type: Superiority; p = 0.0056, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.00002, 95% CI 2-sided [-1 to -0.00002] — Lower is better

ADVERSE EVENTS:
Time Frame: During the study (12 weeks).
Description: Adverse/Serious adverse events were registered in patients of the Safety population (n=390).
Groups:
- Placebo-2 + Placebo-4: Placebo-2 (2 tablets twice daily) and Placebo-4 (2 tablets 4 times daily)
  Raw data from groups placebo-2 and placebo-4 was pooled into combined Placebo group. In accordance with study protocol no dose dependency in placebo effect was assumed. In accordance with study protocol no regiment dependency in placebo effect was assumed.
Arm/Group | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) | Placebo-2 + Placebo-4
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/131 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/131 | 0/132
Other Adverse Events (participants affected / at risk) | 8/127 | 12/131 | 17/132
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenoten, 2 Tablets Twice Daily (4 Tablets/Day) (N=127) | Tenoten, 2 Tablets 4 Times Daily (8 Tablets/Day) (N=131) | Placebo-2 + Placebo-4 (N=132)
Palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Retinal angiopathy
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Vaginosis bacterial NOS
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Acute tonsillitis
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Periorbital contusion
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Lumbar pain
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Cramps in legs (calf)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Osteochondrosis of spine
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Taste metallic
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4) — Headache NOS, temporal headache, headache unilateral, headache fullness
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) — Daytime sleepiness, sleepiness
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03036293/Prot_SAP_000.pdf